CLINICAL TRIAL: NCT07312955
Title: Efficacy of Combination of Solifenacin and Tadalafil Versus Solifenacin Alone in Treatment of Overactive Bladder in Females
Brief Title: Solifenacin Plus Tadalafil vs Solifenacin Alone for Overactive Bladder in Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Sabbah, Resident of Urology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MS 386/2025
Record Dates: First submitted 2025-12-16; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Overactive Bladder
Keywords: Overactive bladder; Urinary urgency; Urinary frequency; Nocturia; Urge urinary incontinence; Solifenacin; Tadalafil; Antimuscarinic agents; Phosphodiesterase 5 inhibitors; Overactive Bladder Symptom Score; Women; Females
MeSH Terms: conditions — Urinary Bladder, Overactive; Nocturia; Urinary Incontinence, Urge | interventions — Solifenacin Succinate; Tadalafil

STUDY DESIGN:
Intervention Model Description: Participants are randomized 1:1 to receive solifenacin 5 mg alone or solifenacin 5 mg plus tadalafil 5 mg for 3 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Solifenacin 5 mg Alone (Active Comparator): Solifenacin (oral tablet) 5 mg once daily for 3 months.
  Interventions: Drug: Solifenacin
- Solifenacin 5 mg + Tadalafil 5 mg (Experimental): Solifenacin (oral tablet) 5 mg once daily plus tadalafil (oral tablet) 5 mg once daily for 3 months.
  Interventions: Drug: Tadalafil

INTERVENTIONS:
Drug: Solifenacin — Solifenacin 5 mg oral tablet, once daily for 3 months.
  Arms: Solifenacin 5 mg Alone
Drug: Tadalafil — Tadalafil 5 mg oral tablet, once daily for 3 months.
  Arms: Solifenacin 5 mg + Tadalafil 5 mg

SUMMARY:
Overactive bladder (OAB) is characterized by urinary urgency with or without urge urinary incontinence, usually with frequency and nocturia, in the absence of urinary tract infection or other obvious pathology. Antimuscarinic agents such as solifenacin are commonly used but may provide incomplete symptom control. Tadalafil (a Phosphodiesterase type 5 inhibitorsinhibitor) has been reported to improve lower urinary tract symptoms and may offer additional benefit in overactive bladder. This randomized controlled trial evaluates the efficacy and tolerability of solifenacin 5 mg plus tadalafil 5 mg versus solifenacin 5 mg alone in females with overactive bladder using the Overactive Bladder Symptom Score (OABSS).

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18 to 60 years.
* Symptoms of overactive bladder for more than 6 months.
* Not receiving current medical treatment for overactive bladder.
* Normal liver function tests.
* Normal kidney function.

Exclusion Criteria:

* Congestive heart failure or history of recent cardiovascular events.
* Currently on medical treatment for overactive bladder.
* Urinary tract infection (eligible only after treatment and resolution).
* Urinary bladder stones.
* Post-void residual urine > 100 cubic centimeter (cm³).
* Closed-angle glaucoma or recent ocular problems.
* Postural hypotension.
* History of neurological disorders (e.g., parkinsonism).
* History of intestinal obstruction.
* Pregnancy or planning pregnancy.
* Myasthenia gravis.
* Severe hepatic impairment.
* History of hypersensitivity to solifenacin or tadalafil.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-11-15 (Actual); Study Completion 2025-11-15 (Actual)

PRIMARY OUTCOMES:
Change in total Overactive Bladder Symptom Score (OABSS) at 1 month | Baseline and 1 month
  Difference in total OABSS (sum of frequency, nocturia, urgency, and urge incontinence domain scores; higher scores indicate worse symptoms) from baseline to 1 month.

SECONDARY OUTCOMES:
Change in total Overactive Bladder Symptom Score (OABSS) at 3 months | Baseline and 3 months
  Difference in total OABSS from baseline to 3 months.
Incidence of adverse effects (tolerability) | Up to 3 months
  Number and percentage of participants reporting adverse effects during the treatment period.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospital (Urology Department), Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the reported results (including OABSS total and domain scores and adverse event data) and a data dictionary will be made available to qualified researchers upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning after publication of the primary results (or thesis acceptance) and available for (e.g., 5 years).
Access Criteria: Requests should include a brief proposal and analysis plan. Access will be provided after review and approval by the study investigators/department and execution of a data use agreement. Data will be shared in a secure format.